CLINICAL TRIAL: NCT01224561
Title: Adaptation of Lipid and Energy Metabolism During a Lipid Overnutrition in Constitutional Thinness
Acronym: Surnutrition
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Clément CAILLAUX, Centre Hospitalier Universitaire de Saint-Etienne
Other Study IDs: 0701047; 2007-A00744-49 (Other: Afssaps); DGS2007-0536 (Other: DGS)
Record Dates: First submitted 2010-10-18; First posted 2010-10-20 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2011-05

CONDITIONS: Lipid Overnutrition; Constitutional Thinness
Keywords: Thinness; Leanness; healthy volunteers; Lipid metabolism disorder
MeSH Terms: conditions — Thinness; Lipid Metabolism Disorders

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — muscle tissue fat tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Constitutional thinness: Women with a a body mass index of less than 16.5 kg/m2
  Interventions: Behavioral: Lipid overnutrition
- Healthy Volonteer: Women with a body mass index between 20 and 25 kg/m2
  Interventions: Behavioral: Lipid overnutrition

INTERVENTIONS:
Behavioral: Lipid overnutrition — During 4 months, the daily caloric intake will be increased by about 70 g fat as butter 20 grams, 100 grams of cheese (Emmental) and 40 grams of almonds. This overnutrition corresponds to an excess of 760 kcal / day or 21,280 calories for the period and then taken to a theoretical 2.4 kg of fat (1 kg fat = 9000 kcal).

SUMMARY:
For a given food intake, fat and energy metabolism in adipose tissue and muscle adapt to nutrient intakes. This adaptation to nutrition may be impaired in susceptible individuals or in obese patients by promoting weight gain, either in constitutional thinness (MC) by blocking it. The MC is a little known entity. These patients wish to grow for her and others. Can they? We have demonstrated abnormalities of hormones regulating appetite (ghrelin, PYY, GLP1 and leptin) that may participate in thinness. Furthermore, this thinness is associated with osteoporosis in 25% of true MC who is 25 years old.

DETAILED DESCRIPTION:
This project aims to overfed MCs and follow the control parameters of energy metabolism. We will look for abnormalities in the adaptation to overnutrition in subjects with genetic background of thinness, which could explain the resistance to weight gain. The answer could possibly help to understand obesity.

ELIGIBILITY:
Inclusion Criteria:

* consent form the study signed
* consent form for genetic study signed
* normal laboratory values for liver enzymes, glucose, lipid

Exclusion Criteria (common to the two groups):

* pregnant
* vegetarian
* heavy smoking
* heavy alcohol
* depressive
* taking hypolipidemic or antihypertensive drugs
* dyslipidemia

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Constitutionnal thinness women and healthy volonteers(women)
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2008-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
gene expression | After one month of lipid overnutrition
  Level of genes (which regulate the lipid and energy metabolism) expression in fat and muscle tissues

SECONDARY OUTCOMES:
Anthropometric parameter | After one month of lipid overnutrition
  Lean mass
Autonomic nervous system activity | After one month of lipid overnutrition
  Heart rate variability analyses using ECG Holter monitoring
gastrointestinal hormone level | After one month of lipid overnutrition
  Serum level of GLP1
Anthropometric parameter | After one month of lipid overnutrition
  Weight
Anthropometric parameter | After one month of lipid overnutrition
  Fat mass
gastrointestinal hormone level | After one month of lipid overnutrition
  Serum level of ghréline
gastrointestinal hormone level | After one month of lipid overnutrition
  Serum level of PYY

CONTACTS AND LOCATIONS:
Overall Officials: Bruno ESTOUR, MD PhD, Principal Investigator — CHU de Saint-Etienne
Locations (3):
- France (3):
  - CRNH Auvergne, Clermont-Ferrand
  - CRNH Rhône-Alpes, Lyon
  - CHU de Saint-Etienne, Saint-Etienne